CLINICAL TRIAL: NCT04535765
Title: Effect of Early Warm Water Sitz Bath on Urinary Retention After Hemorrhoidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cathay General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CGH-P108094
Record Dates: First submitted 2020-06-14; First posted 2020-09-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Hemorrhoids; Haemorrhoids; Piles; Hemorrhoidal Disease
Keywords: hemorrhoidectomy; warm water sitz bath; urinary retention
MeSH Terms: conditions — Hemorrhoids; Urinary Retention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The experimental group began to perform warm water sitz bath 6 hours after the operation (the day of the operation).Warm water sitz bath temperature is 41-43 ℃, 3 times a day, 5 minutes each time.
  Interventions: Other: early warm water sitz bath
- control group (Other): The control group began to perform warm water sitz bath at 8:00 in the morning on the first day after the operation as usual.Warm water sitz bath temperature is 41-43 ℃, 3 times a day, 5 minutes each time.
  Interventions: Other: Regular time warm water sitz bath

INTERVENTIONS:
Other: early warm water sitz bath — The experimental group started the warm water sitz bath 6 hours after the end of the hemorrhoid surgery.
  Arms: experimental group
Other: Regular time warm water sitz bath — According to the routine, the control group started the warm water sitz bath on the first day after the hemorrhoid surgery.
  Arms: control group

SUMMARY:
Background:

Hemorrhoid is one of the most common chronic anorectal diseases. The prevalence rate is about 44%. It occurs in adults aged 45-65 years. Hemorrhoidetomy resection is still the standard treatment for grade III and IV hemorrhoid. Urinary retention is one of the most common complications after hemorrhoid surgery, and the complications occur within 24 hours after surgery. The warm water sitz bath is a routine nursing care after hemorrhoid surgery in the clinic. The purpose is to provide moist heat of the perineum and anus to clean, promote healing and drainage, relieve pain, stimulate urination and promote relaxation. In contrast, all current studies, warm water sitz bath intervention time is the first day after surgery, the complications within 24 hours after surgery are not alleviated.

Objective:

The main purpose was to use experimental research methods to verify the effect of early warm water sitz bath on urinary retention after hemorrhoidectomy. The secondary objective was the effect of early warm water sitz bath on wound pain after hemorrhoidectomy.

Methods:

This study was a single-blind randomized trial in which subjects were randomly assigned to an experimental or control group with symptomatic stage III or IV end hemorrhoid who were admitted to the hospital for hemorrhoidectomy. The experimental group started the warm water bath 6 hours after the end of the operation, while the control group started the warm water sitz bath on the first day after the operation. The investigator assessed the amount of residual urine and wound pain index before and after each operation of the warm water sitz bath after surgery, and each subject was evaluated 8 times until 24 hours after surgery.

DETAILED DESCRIPTION:
In order to ensure that the results of the study are not distorted by humans, this study is a single-blind randomized trial study. The subjects were randomly assigned to the experimental group or the control group with a permuted block randomization. For the sample number calculation, refer to Hedeker, Gibbons & Waternaux (1999) Comparing the time-dependent comparison of the longitudinal design sample size estimates between the two groups, and considering the 20% sample loss rate, the total number of samples is estimated to be 64 (32 in the control group and 32 in the experimental group).

The two groups of patients also received the same conventional treatment, anesthesia and surgery on the night before and on the day of the operation, and the warm water sitz bath was performed at different times after the operation. The warm water sitz bath temperature of the two groups was also 41-43°C daily 3 times (9:00, 13:00, 17:00), 5 minutes each time, and regularly take the same painkillers, stool softeners, and antibiotics. The researchers evaluated the wound pain index on the Numerical Rating Scale (NRS) 6 hours after the operation, 7 hours after the operation, and before and after each warm water sitz bath; After urine, the residual urine volume of the subject was evaluated with a Bladder Scan until the first day after the operation. A total of 8 evaluations were performed: 6 hours after the operation, 7 hours after the operation, and the first day after the operation 8:30, 9:30, 12:30, 13:30, 16:30, 17:30.

During the test, the number of subjects with adverse reactions (vertigo, weakness, sustained wound bleeding greater than 100ml) was greater than 3% of the total number of cases (2 persons). The trial was terminated immediately.

Acceptance conditions:

1. Age over 20 years old, easy to move, can get out of bed and take a bath.
2. Symptomatic grade III or IV hemorrhoids diagnosed by the surgeon.
3. Accept epidural anesthesia.
4. Perform hemorrhoidectomy.
5. Those who have clear awareness and are willing to participate in and fill out the research consent form.

Exclusion conditions:

1. Diseases around the anus (fistula, abscess).
2. Urinary tract problems (prostate hypertrophy in the past medical history; urinary tract infections on admission routine urine tests, urinary retention as assessed by Bladder Scan).
3. Take painkillers before surgery.

Statistical methods

1. Descriptive statistical analysis: Adopt the mean, standard deviation, frequency distribution and percentage to present the basic attributes of the subjects.
2. Inferential statistics: Chi-square test was used to analyze the categorical variables, and independent sample t-test was used to analyze the continuous variables.
3. Use the independent sample t test to compare the differences in the average degree of urinary retention and pain between the groups. If the data are not normally distributed, switch to the Mann-Whitney U test without parental analysis to compare the experimental group and the control group before and after bathing Whether there is a difference, p value <0.05 is considered statistically significant.
4. Use GEE (Generalized Estimating Equation) to check whether there is any difference in the degree of urinary retention and pain in each group.

The use of k-Nearest Neighbours to fill in the missing values is mainly to see that the relevant data measured by the subject in the same group is similar to those of other subjects, and then average the data measured by these similar subjects at the same time Value to fill.

ELIGIBILITY:
Inclusion Criteria:

1. The age is more than 20 years old, the action is convenient, you can get out of bed and take a bath.
2. Diagnosed as symptomatic grade III or IV hemorrhoid by a surgeon.
3. Accept epidural anesthesia.
4. Perform an open hemorrhoidectomy.
5. After the researcher explains the purpose of the study, the person with a clear consciousness and willing to participate and fill out the study consent form.

Exclusion Criteria:

1. Disease around the anus (fistula, abscess).
2. Urinary tract problems (in the past, there was a hypertrophy of the prostate; the routine urine test for admission had a urinary tract infection, and the bladder volume tester evaluated urinary retention).
3. Take analgesics before surgery.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Effect of early warm water sitz bath on urinary retention after hemorrhoidectomy | In this study, a Bladder Scan was used to evaluate the residual urine volume 6 hours after the operation, 7 hours after the operation and before and after each warm water sitz bath, a total of 8 times.
  The main purpose was to use experimental research methods to verify the effect of early warm water sitz bath on urinary retention after hemorrhoidectomy.This study is expected to use the bladder scan BVI 6100 as a tool for evaluating urinary retention. It is currently used clinically to measure bladder urine volume. Studies have indicated its accuracy, sensitivity, and specificity, with results of 94%, 97%, and 91%, respectively (Attia, Hiligsmann, Hellinckx, Wijnen & Evers, 2016).
  Before investigating the receipt, the researcher must go through three bladder volume tester operation tests and measure the bladder urine volume in accordance with the standard procedures of the instrument operation. Measurement of residual urine volume.

SECONDARY OUTCOMES:
Effect of early warm water sitz bath on wound pain after hemorrhoidectomy | In this study, the wound pain index was evaluated with a Numerical Rating Scale (NRS) 6 hours after the operation, 7 hours after the operation, and before and after each warm water sitz bath, a total of 8 times.
  The secondary objective was the effect of early warm water sitz bath on wound pain after hemorrhoidectomy.This study used a Numerical Rating Scale (NRS) to assess wound pain after hemorrhoidectomy. NRS is the most suitable pain scale for patients after surgery. The patient evaluates his pain on a scale of 0 to 10, where 0 means no pain; 1-3 mild pain; 4-6 moderate pain; 7-10 severe pain ( Karcioglu et al., 2018; Aryolcu, 2014). Li et al. (2007) studied the reliability and validity of the NRS scale and the quantification scale. The results showed that the current (current) pain, the most severe (worst) pain, the least (least) pain and the average (average) pain The reliability of ICC (Interclass correlation coefficient) is .822.

CONTACTS AND LOCATIONS:
Locations (1):
- Cathay General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liao WC, Cheng YY, Hsu CK, Chiu YC, Chiu HY, Chang SC, Hu SH. Effects of early warm water sitz bath on urinary retention and pain after haemorrhoidectomy: A randomized controlled trial. Int J Nurs Stud. 2024 Jun;154:104765. doi: 10.1016/j.ijnurstu.2024.104765. Epub 2024 Mar 31. PMID 38642473